CLINICAL TRIAL: NCT05982548
Title: The Use of a Virtual Reality Intervention on Stigma, Empathy and Attitudes Towards People With Psychotic Disorders Among Mental Healthcare Professionals
Brief Title: The Use of a Virtual Reality Intervention on Stigma, Empathy and Attitudes Towards People With Psychotic Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Mental Health, Singapore (Other)
Responsible Party: Principal Investigator, Tay Jing Ling, Advanced Practice Nurse, Institute of Mental Health, Singapore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2023/00027
Record Dates: First submitted 2023-07-24; First posted 2023-08-08 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Mental Disorder
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The VR intervention was created using the Unreal Engine software (Unreal Engine, 2022). The VR intervention includes the scenario of a home.
  Participants will view the home as a first person character and experience psychotic phenomena including auditory hallucinations. The intervention will be delivered in one setting and lasts no more than seven minutes. It will be disseminated using smartphone inserted into VR headset equivalent of google cardboard.
  Interventions: Other: VR intervention
- VR control group (Active Comparator): The VR control group will view the scenario of the same home without the simulated visual and auditory hallucinations.
  Interventions: Other: VR control intervention

INTERVENTIONS:
Other: VR intervention — VR intervention of no more than 7 minutes
  Participants viewed the home as a first person character and experience psychotic phenomena including auditory hallucinations.
  Arms: Intervention group
Other: VR control intervention — VR intervention of no more than 7 minutes
  Participants viewed the same home as a first person character without psychotic phenomena
  Arms: VR control group

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of a VR intervention on (1) stigma, (2) empathy and (3) attitudes towards those experiencing mental disorders.

Participants will review a VR intervention, and complete questionnaires at pre-test, post-test and one month follow-up.

Researchers will compare the VR intervention with a control VR intervention to evaluate the varying effects on stigma, empathy and attitudes towards those experiencing mental disorders.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are aged at least 21 years old
* Employed by the Institute of Mental Health as a physician, allied health professional or nurse.
* understands English
* work directly with patients.

Exclusion Criteria:

* unable to use virtual reality interventions due to reasons including motion sickness, disorientation, nausea and vomiting.
* history of epilepsy

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-07-17 (Estimated); Study Completion 2024-07-17 (Estimated)

PRIMARY OUTCOMES:
Desire for Social Distance | pre-intervention, immediately after the intervention, follow-up at 1 month after intervention
  Desire for Social Distance Scale
  The eight questions are rated on a four-point Likert scale:
  yes, definitely (0), yes, probably (1), probably not (2) and definitely not (3) with greater scores implying greater desire for social distancing.
Personal Stigma | pre-intervention, immediately after the intervention, follow-up at 1 month after intervention
  Personal Stigma Scale Personal Stigma Scale consisted of two subscales: 'Personal unpredictable/ dangerousness' and 'Personal weak not sick' The questions were calculated as 'strongly agree' (4) to 'strongly disagree' (0), with greater scores implying greater stigmatizing attitudes.
Empathy | pre-intervention, immediately after the intervention, follow-up at 1 month after intervention
  Empathetic concern sub-scale of Interpersonal Reactivity Index The 7-item sub-scale is measured on a five point likert scale ranging from 'does not describe me well' (0) to 'describes me very well' (4).
Attitudes towards those experiencing mental disorders | pre-intervention, immediately after the intervention, follow-up at 1 month after intervention
  modified Attitudes Towards People with Schizophrenia scale The 7-item scale is measured on a nine point likert scale ranging from (1) to (9). Greater scores equate better attitude towards people with schizophrenia.

SECONDARY OUTCOMES:
Demographic data | pre-intervention
  occupation, gender, marital status, ethnic groups, age, years of service
Acceptability of the intervention | immediately after the intervention
  Authors constructed questionnaire to assess for acceptability of intervention. A total of 10 questions consisting of 6 multiple choice questions ranging from strongly disagree to strongly agree on a 7-point likert scale. An example of one question is, 'I find the intervention engaging'.
  It also consists of 4 open ended questions. Example of one question is, 'Please list the strength of the intervention'
Safety of VR intervention | immediately after the intervention
  Visually induced motion sickness susceptibility questionnaire:
  It consists of six questions that evaluates presence of adverse effects from using the VR intervention from 'never' (0) to 'often' (3).

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Mental Health, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tay JL, Qu Y, Lim L, Puthran R, Tan CLR, Rajendran R, Wei KC, Xie H, Sim K. Impact of a Virtual Reality Intervention on Stigma, Empathy, and Attitudes Toward Patients With Psychotic Disorders Among Mental Health Care Professionals: Randomized Controlled Trial. JMIR Ment Health. 2025 Jan 21;12:e66925. doi: 10.2196/66925. PMID 39836956